CLINICAL TRIAL: NCT06779331
Title: Phosphate Urine Excretion in Critically Ill Patients - a Prospective Observational Study
Brief Title: Phosphate Urine Excretion in Critically Ill Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Liran Statlender, physician, Rabin Medical Center
Other Study IDs: RMC-0149-23
Record Dates: First submitted 2025-01-08; First posted 2025-01-16 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Critically Ill Intensive Care Unit Patients
Keywords: phosphate; hypophosphatemia; hyperphosphatemia; urine collection
MeSH Terms: conditions — Hypophosphatemia; Hyperphosphatemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- early hypophosphatemia: patients who developed first hypophosphatemia (Pi<2.5mg/dL) within 24 hours of ICU admission
- hypophosphatemia: patients who developed first hypophosphatemia (Pi<2.5mg/dL) at least 24 hours after ICU admission, within study observation period
- Normophosphatemia: patients who did not develop neither hypophosphatemia (Pi<2.5mg/dL) nor hyperphosphatemia (Pi>4.5mg/dL) during study observation period.
- Hyperphosphatemia: patients who developed hyperphosphatemia (Pi>4.5mg/dL) during study observation period.

SUMMARY:
Hypophosphatemia is a common disorder in critically ill patients, appearing in 15-35% of Intensive Care Unit (ICU) admissions. Its reasons are multifactorial, including sepsis, refeeding syndrome, and continuous renal replacement therapy. Hypophosphatemia is generally accepted as a predictor of poor outcomes, such as prolonged ventilation and higher mortality. However, conflicting evidence exists and several works demonstrated no effect on length of ventilation, nor mortality. We have recently demonstrated no effect of hypophosphatemia on mortality and length of ventilation. However, both parameters were affected by energy delivery to the patient, with higher energy delivery associated with lower mortality and longer length of ventilation, suggesting a complex interaction between energy delivery to the patient, hypophosphatemia appearance, and patient outcomes. This raised hypothesis that hypophosphatemia is a marker of recovery, as in fulminant hepatic failure, or recovery after hepatectomy.

Phosphate is mainly an intracellular anion, with only 1% of its total body amount is extracellular. It is absorbed from the small intestine, mainly at the jejunum, both through passive para-cellular and active trans-cellular process. Phosphate is excreted in the urine, after being filtered in the glomeruli, and reabsorbed mainly in the proximal tubule (less than 10% of the reabsorption occurs in the distal nephron), by sodium-phosphate co-transporters. Phosphate regulation in the body is complex. It is regulated by vitamin D, parathyroid hormone (PTH), and fibroblast growth factor 23 (FGF-23). Therefore, phosphate regulation is affected both from intestine dysfunction and kidney injury. Although hyperphosphatemia in various kidney injury is well described, the effect of kidney function regarding phosphate excretion in critically ill patients with hypophosphatemia has been scarcely described. French and Bellomo described 7 patients who had decreased phosphate kidney reabsorption during hypophosphatemia. Charrone et. al demonstrated increased phosphate excretion after IV phosphate infusion to 47 critically ill patients with hypophosphatemia. Dickerson et. al demonstrated higher rates of hypophosphatemia in 20 thermally injured patients (compared to 20 multiple trauma patients) despite greater phosphate delivery through nutrition, along with increased (although insignificant) phosphate urinary excretion in this group. This might suggest that increased renal phosphate loss has a role in hypophosphatemia development. Better understanding these processes is important, with regard to the effect of nutritional support and hypophosphatemia effects on patients' outcomes. This study aims to describe urinary phosphate excretion in critically ill patients with regard to kidney function, phosphate serum level, and phosphate intake.

DETAILED DESCRIPTION:
Data collection

We will document the following data for each patient, for maximum of five days from admission:

* Demographic data, including age; sex, height, weight, admission reason to ICU.
* Acute Physiology And Chronic Health Evaluation II (APACHE II) Score (24 hours after ICU admission)
* Daily Sequential Organ Failure Assessment (SOFA) Score and SOFA components.
* Daily Ventilation status
* Daily vasopressor requirement
* Daily Renal replacement therapy (if any)
* Daily urine volume
* Daily fluid balance - including daily fluid input and output
* Daily 6 hours urine collection, with documentation of collection volume, urine creatinine, and urine electrolytes. Specimens from the first two days of admission will be sent to laboratory analysis only after the patient is admitted for more than 48 hours.
* Calculation of glomerular filtration rate (GFR) based on urine collection findings.
* Calculation of phosphate excretion amount based on urine collection findings - both maximal phosphate tubular reabsorption rate (TmP) and Fractional Excretion of phosphate (FePi).
* Daily serum phosphate and calcium levels
* Daily phosphate intake - from enteral nutrition, parenteral nutrition, and supplemental (enteral and parenteral).
* For the last 60 patients - a single measurement of PTH and vitamin D.
* Patient outcomes: ICU length of stay; Hospital length of stay; Length of ventilation; Ventilator free days at 28 days; Mortality - at ICU, during hospital admission, and at 28 & 90 days.

ELIGIBILITY:
Inclusion Criteria:

Adult (>18) Critically ill patients who are admitted for at least 48 hours in the ICU, who are being ventilated in the first time it's 00:00 during their admission, with a urinary foley catheter.

Exclusion Criteria:

* Age < 18 years
* Pregnancy.
* Recent admission to an ICU (within 30 days)
* Chronic kidney disease treated with hemodialysis.
* Oral nutrition by the patient at admission time
* Existence of another urinary catheter (e.g nephrostomy), or ileal conduit.
* Hematuria
* RRT treatment within 48 hours of admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients who were admitted to the ICU
Sampling Method: Non-Probability Sample
Enrollment: 205 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
90 day mortality | 90 days from ICU admission
  Mortality within 90 days of ICU admission.

SECONDARY OUTCOMES:
28-Ventilation free days | 28 days of ICU admission
  Number of ventilator free days within 28 days of ICU admission
ICU Length of stay | 90 days from ICU admissino
  ICU admission duration
hospital length of stay | up to 90 days after ICU admission
  hospital admission duration
ICU and hospital mortality | 90 days from ICU admissino
  whether mortality happened during ICU/hospital admissino
Differences in Glomerular Filtration Rate | Daily during first five days of ICU admission
  Differences in glomerular filtration rate (GFR) (ml/min)
Maximal tubular reabsorption of phosphate (TmP) | Daily during first five days of ICU admission
  Differences in Maximal tubular reabsorption of phosphate (TmP) (mg/min) will be examined in each group and between groups.
Phosphate Balance | Daily during first five days of ICU admission
  Differences in phosphate balance (mg) will be examined between the groups
Ratio of Maximal Tubular Reabsorption rate to Glomerular Filtartaion Rate (Tmp/GFR) | Daily during first five days of ICU admission
  Differences in the ratio Tmp/GFR (mg/ml), and daily phosphate balance will be examined in each group and between groups.
PTH level and Vitamin D level | One measurement, during first five days of ICU admission
  Differences in PTH (ng/ml) and Vitamin D (IU/ml) between groups
caloric intake | daily measurement during first five days of ICU admission
  Differences in the caloric intake provided (Kcal/day) will be examined between the groups
timing of nutritional support initiation | within first five days of ICU admission
  timing of nutritional support initiation will be compared between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medcial Center, Petah Tikva, Israel